CLINICAL TRIAL: NCT05741320
Title: Are Anesthetists Still Secret Heroes After the Pandemic?
Brief Title: Anesthetists After the Pandemic in the Eyes of the Public
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Aygun cuhadar, anesthesiology and reanimation md, Ankara City Hospital Bilkent
Other Study IDs: E1-21-2118
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Anesthesia; COVID-19 Pandemic
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- public: Subjects older than 16 years of age and not working in any health sector will be included in the study.
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — 27 questions will be asked to public to find out what is the role of anesthetists after the covıd pandemic

SUMMARY:
Anaesthesia and anesthesiologist from the very beginning has obtained "Behind the screen" role. This is of great concern as the field of Anesthesiology has expanded its services to various specialities like intensive care, postoperative pain management, labour analgesia, accident and trauma management, casualty etc. the role assigned to the anesthesiologist remains inaccurate even during COVID 19 pandemic.

The aim of this study was to evaluate general publics' perception about anesthesiologist& anesthesia in operating and especially intensive care units during COVID 19 pandemic.

DETAILED DESCRIPTION:
Method: A questionnaire consisting of 27 questions was asked to fill by the general population via the social media. The questionnaire consists of two parts: The first part includes demographic data such as age, gender, education level, occupation; the second part includes the questions about anesthesia experience and knowledge.

ELIGIBILITY:
Inclusion Criteria:

- Subjects older than 16 years of age and not working in any health sector will be included in the study.

Exclusion Criteria:

* if she/he doesn't want to join

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects older than 16 years of age and not working in any health sector will be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
who are the anesthesist | questionare will be administered online for a one month period.
  the anesthetist's role will be evaluated by yes-no or don't know
covid19 and anesthetists | questionare will be administered online for a one month period.
  Whether anesthetists' duties during the covid19 pandemic are known to the public will be evaluated with yes, no or I don't know.

CONTACTS AND LOCATIONS:
Locations (1):
- Aygün Güler, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Swinhoe CF, Groves ER. Patients' knowledge of anaesthetic practice and the role of anaesthetists. Anaesthesia. 1994 Feb;49(2):165-6. doi: 10.1111/j.1365-2044.1994.tb03380.x. PMID 8093141
- [Background] Whitty P, Goodwin D, Shaw IH. Patients' perception of the anaesthetist and anaesthesia. Anaesthesia. 1994 Jul;49(7):644-5. doi: 10.1111/j.1365-2044.1994.tb14248.x. No abstract available. PMID 8042743
- [Background] van Klei WA, Hollmann MW, Sneyd JR. The value of anaesthesiologists in the COVID-19 pandemic: a model for our future practice? Br J Anaesth. 2020 Nov;125(5):652-655. doi: 10.1016/j.bja.2020.08.014. Epub 2020 Aug 20. No abstract available. PMID 32896431
- [Background] Ribeiro CS, Mourao JI. Anesthesiologist: the patient's perception. Braz J Anesthesiol. 2015 Nov-Dec;65(6):497-503. doi: 10.1016/j.bjane.2014.05.014. Epub 2015 Sep 28. PMID 26614148
- [Background] Onutu AH, Rus C, Acalovschi I. The public perception of the anaesthesiologist in Romania: a survey. Rom J Anaesth Intensive Care. 2017 Apr;24(1):21-28. doi: 10.21454/rjaic.7518.241.onu. PMID 28913494
- [Background] Sagun A, Birbicer H, Yapici G. Patients', who applied to the anesthesia clinic, perceptions and knowledge about anesthesia in Turkiye. Saudi J Anaesth. 2013 Apr;7(2):170-4. doi: 10.4103/1658-354X.114076. PMID 23956718